CLINICAL TRIAL: NCT06775509
Title: Optical Quality of the Cornea in Orthokeratology
Acronym: COPCORTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Jose Licari, Ophtalmologist Doctor, Institut Investigacio Sanitaria Pere Virgili
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27-09-23v1
Record Dates: First submitted 2024-12-11; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Myopia (Disorder); Astigmatism
Keywords: Ortho-K; Overnight Orthokeratology; Progression of Myopia; Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Masking Description: Statistical Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ortho - k (Experimental): The Utilization of Otho-K Contact lenses
  Interventions: Device: Ortho-K

INTERVENTIONS:
Device: Ortho-K — Utilization of Ortho-K Contact Lenses for The Treatment of Myopia

SUMMARY:
Analyzing Optical Quality After the Use of Overnight Orthokeratology (Ortho-K)

DETAILED DESCRIPTION:
Optical Quality of the Cornea in Orthokeratology

Influence of changes in total corneal refractive power, corneal asphericity, and epithelial thickness.

Introduction:

The cornea is the transparent and avascular tissue of the eye, consisting of five layers: the corneal epithelium, Bowman's membrane, the stroma, Descemet's membrane, and the endothelium. Its thickness varies, being thinner at the central level, approximately 520 microns (0.52 mm), and about 1 mm near the sclera.

The corneal epithelium, the outermost layer, not only provides strong protective functions but also plays a role in corneal refractive function. In particular, the central corneal epithelium is especially important for corneal refraction. The refractive action of any optical surface is governed by two main parameters: the curvature of its surface and the difference in refractive indices of the media it separates.

Unlike other ocular media, the cornea is considered a refractive surface, as most refraction occurs at its anterior surface. This is due to the significant difference in the refractive index between air (n=1) and the corneal interior (n=1.376), which provides a refractive power of approximately 49 diopters. The posterior surface of the cornea, on the other hand, separates two media with very similar indices; the aqueous humor (n=1.336) has a slightly lower index than the cornea, reducing the overall refractive power of the cornea to about 43 diopters.

Asphericity is a characteristic of the cornea, with the central part being more curved than the peripheral zone. The Q value measures the corneal asphericity index (Q = 0 for spherical corneas, Q < 0 for prolate corneas, and Q > 0 for oblate corneas). The human cornea typically has a prolate shape (average negative Q value of - 0.27).

The Q value is based on a central curvature of 3 to 4 mm of the cornea. It is a coefficient that describes the rate of curvature change from the center to the periphery based on corneal radius values. The normal shape of the cornea is not a sphere but a prolate ellipse, meaning its curvature flattens as movement occurs from the center to the periphery. Prolate corneas, which are flatter in the periphery (negative Q values), reduce spherical aberrations due to their curvature. Conversely, oblate corneas, with positive Q values and a more curved periphery than the central part, increase spherical aberrations.

Orthokeratology (Ortho-K) is a clinical technique that temporarily reshapes the cornea to eliminate or reduce refractive errors. Ortho-K lenses are commonly worn during sleep (overnight orthokeratology) and removed immediately upon waking, allowing clear vision without assistance throughout the day. These lenses are made of rigid gas-permeable (RGP) material and aim to reduce myopia by flattening the cornea. This treatment is reversible, safe, and FDA-approved.

Although orthokeratology reduces myopia and provides good uncorrected vision during the day, numerous studies have shown that the combination of central corneal flattening and mid-peripheral corneal thickening leads to a significant increase in higher-order aberrations, resulting in a decrease in visual quality.

From a more physical perspective, light can be defined as an electromagnetic wave characterized by a wavefront. A wavefront is the surface where all points of the medium are reached by the wave at the same time. It is inferred that the wavefront is the surface formed by all points with the same phase as the wave propagates. The direction of a ray is always perpendicular to the wavefront.

The term aberration refers to deviation or distortion. Any alteration or change in the wavefront as it passes through an optical medium (ocular or otherwise) causes non-ideal propagation, resulting in wavefront aberration. The difference between the ideal and aberrated paths is known as wavefront aberration or wavefront error. Wavefront aberrations can be described using Zernike polynomials to specify ocular aberrations, allowing any aberration to be expressed in this way.

With orthokeratology, higher-order corneal aberrations increase significantly, especially spherical aberration. These increases correlate with the degree of myopic correction. Several studies have concluded that the loss of optical quality is most noticeable within the first month and becomes insignificant in subsequent months. After short-term corneal reshaping, optical quality decreases to a certain degree, but the loss is acceptable.

As mentioned earlier, orthokeratology causes central corneal epithelial thinning and mid-peripheral epithelial thickening. Changes in epithelial thickness show a non-uniform pattern, with greater thinning in the temporal and inferior zones compared to the nasal and superior zones in the paracentral region, and greater thickening in the nasal zone compared to the temporal zone in the mid-periphery.

Main Objective:

To analyze the optical quality of the cornea after changes induced in its shape and structure by overnight orthokeratology.

To achieve this, the following will be analyzed:

Changes in the various refractive maps obtained using the Pentacam topography system.

Corneal aberrations obtained through Zernike analysis of both corneal surfaces. The changes in the anterior corneal asphericity and its correlation with induced spherical aberration will also be analyzed.

Changes in central and peripheral epithelial thickness and their correlation with changes in corneal asphericity and induced aberrations evaluated using corneal OCT.

Changes in the aforementioned variables between morning and late afternoon (daily regression).

In all cases, the results will also be correlated with ocular refraction obtained under cycloplegia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 8 and 21 years old. Those who accept to participate in the study. The use of Ortho-K lenses for 8 to 10 hours per night, once the risks and benefits of using Ortho-K have been explained.
* Refractive error of myopia between -1.00 and -5.00 diopters (D) with astigmatism of 1.50 D or less, with-the-rule.
* Best-corrected visual acuity of 20/20 or better before treatment.
* Ortho-K lens centered or decentered by no more than 0.5 mm radially, determined by slit-lamp examination.

Exclusion Criteria:

* History of hard contact lens use and contraindications for ocular and systemic Ortho-K, determined by a routine examination.
* Patients who have previously undergone any refractive modulation procedure.
* Patients with any corneal pathology, dry eye, glaucoma, retinal pathology, strabismus, ptosis, amblyopia, history of ocular allergy, or infection.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
OPTICAL QUALITY | 1 month after using Ortho-K
  The primary outcome measure is the change in total corneal higher-order aberrations between baseline and 30 days of orthokeratology lens wear. It will be expressed using Zernike coefficients in microns.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Licari Vision, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No